CLINICAL TRIAL: NCT06875700
Title: Beliefs, Attitudes, and Response to Genetic Testing in Sarcoma Patients
Brief Title: Beliefs, Attitudes, and Response to Genetic Testing in SarcomaPatients
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of New South Wales (Unknown); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: HCI165523; 1P50CA272170-01 (NIH)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LMS Probands: LMS Probands are the first person in a family to be known to have a germline predisposition gene mutation in LMS. A cohort of patients with a histologically confirmed leiomyosarcoma diagnosis will be prospectively recruited from two SPORE prospective biomarker studies.
- Relative of LMS Probands: Relatives to LMS probands will be enrolled in this cohort. Approximately 4 family members per proband will be recruited.

SUMMARY:
Genomic research has shown that a portion of leiomyosarcomas can be attributed to an underlying cancer predisposition syndrome. However, the optimal approach for incorporating germline testing into the care of these patients. This study is assessing the beliefs about the heritability of leiomyosarcoma and other cancer risks, and attitudes towards germline testing among leiomyosarcoma patients.

DETAILED DESCRIPTION:
This is a descriptive study to explore attitudes to genomics and return of genetic information and examine the cognitive and affective impact of receiving germline genetic information among LMS patients and their family members.The present study will aim to do the following:

* Assess leiomyosarcoma (LMS) patients' beliefs and attitudes about the heritability of LMS and their interest in genetic testing.
* Among LMS patients who undergo genetic testing, evaluate the cognitive, affective, and communication outcomes of genetic testing in LMS patients found to have actionable germline germline pathogenic variants (PVs).
* Evaluate family members' beliefs and attitudes about the heritability of reasons for undergoing genetic testing and responses.

Prior studies of cancer patients have found a strong interest in genetic testing so at-risk relatives will have the opportunity to have increased cancer screening or take risk-reducing measures to prevent cancer. However, the genes most strongly associated with LMS are tumor protein 53 (TP53) gene and Retinoblastoma 1 (Rb1) gene. These genes cause risks for cancers that families may be less familiar with and that have less well-established approaches for screening and prevention.

LMS may not be the most significant cancer risk related to the syndrome associated with the PV identified. The finding of risk for other non-LMS cancers may be unexpected and incongruent with the family's experience or focus on the LMS being treated. Screening recommendations for relatives testing positive for these PV will generally be given cancer screening recommendations targeted towards risks for cancers other than LMS.

Patients beginning or in the midst of cancer treatment may be less able to share and effectively communicate about genetic test results to patients. We need to better understand how patients and family members respond to findings to maximize the clinical benefit of this information and support family communication.

LMS patients will be identified by querying the enterprise data warehouse (EDW) and Huntsman Tumor Registry and prospectively by reviewing clinic and tumor board lists.

ELIGIBILITY:
Inclusion LMS Proband

* Actionable germline PV detected in the research context
* Living
* No prior germline testing for this PV
* Able to speak and read English
* Mentally competent
* Age 18 or older

Relative of LMS Proband

* 25-50% chance for having inherited the PV
* No prior germline testing for this PV
* Able to speak and read English
* Mentally competent
* Age 18 or older

Exclusion (both cohorts)

* <18 years
* Unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be Patients with a confirmed or suspected diagnosis of LMS and Relatives of LMS patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Beliefs about the heritability of Leiomyosarcoma | up to 1 day from study enrollment
  This outcome will report the count of participants who self-reported a strong belief in heritability. Participants who responded on a questionnaire that sarcoma is somewhat or highly heritable are considered to have a strong belief in heritability.
  This outcome measure will be assessed on Day 1 of the study.

SECONDARY OUTCOMES:
Interest in germline genetic testing | up to 1 day from study enrollment
  This outcome will report the count of participants who self-reported an interest in germline genetic testing. This will report the number of participants who respond on a baseline questionnaire that they are interested in having a genetic test related to cancer risk.

OTHER OUTCOMES:
Uptake in germline genetic testing | up to 1 day from study enrollment
  This outcome will report the count of participants who proceed with germline genetic testing. Participants will be asked on their baseline questionnaire if they have completed germline genetic testing.
Preferences for receiving information about germline testing | up to 1 day from study enrollment
  This outcome will report the count of participants who self-reported sources for genetic testing information as helpful.
  Participants will rank questions about sources of information from "1 Not helpful at all" to "6 Extremely helpful" on their baseline questionnaire. Participants who reported >5 on this scale are considered to have found the source for genetic testing information as helpful.
  This outcome will assess information presented in tables and graphs and information presented numerically.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IDP will be shared with the University of Michigan Rogel Cancer Center for data analysis.